CLINICAL TRIAL: NCT05046418
Title: A Prospective, Observational, Cohort Study Investigating the Clinical Impact of Hypoallergenic Formulae With Synbiotics in Infants With Cow's Milk Allergy
Brief Title: Synbiotics Cohort Study
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: HAFSYN21
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cows Milk Allergy
Keywords: synbiotics; paediatrics; gut microbiome
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hypoallergenic formula containing synbiotics: Infants (aged <13 months) with cow's milk allergy (CMA) who are prescribed a hypoallergenic formula containing synbiotics as part of usual clinical practice for the dietary management of CMA.
  Interventions: Other: Hypoallergenic formula containing synbiotics

INTERVENTIONS:
Other: Hypoallergenic formula containing synbiotics — An extensively hydrolysed formula containing synbiotics or an amino acid formula containing synbiotics.

SUMMARY:
Observational study exploring the clinical outcomes of infants with cow's milk allergy who are prescribed a hypoallergenic formula containing synbiotics.

DETAILED DESCRIPTION:
A range of clinical outcomes will be collected from the medical records and in-person assessment of 60 fully or partially formula fed infants (aged <13 months) who are prescribed a hypoallergenic formula containing synbiotics as part of usual clinical practice for the dietary management of cow's milk allergy

ELIGIBILITY:
Inclusion Criteria:

* Aged <13 months
* Confirmed or suspected CMA- based on healthcare professional (HCP) judgement
* At baseline, parent(s) must already be exclusively or partially formula feeding their child (with a hypoallergenic or non-hypoallergenic formula) or have already made the decision to start exclusively or partially formula feeding
* Recently prescribed a hypoallergenic formula containing synbiotics

Exclusion Criteria:

* Exclusively breastfed infants
* Primary lactose intolerance
* Enterally fed infants
* Premature infants (born <37 weeks) with a corrected age of less than 1 month
* Infants with contraindications to the use of hyopallergenic formula containing synbiotics
* Major hepatic or renal dysfunction
* Investigator concern around the ability of family to comply with protocol and requirements of study

Ages: 0 Months to 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Exclusively or partially formula fed infants with confirmed or suspected CMA who have been prescribed hypoallergenic formula containing synbiotics for the management of CMA as part of clinical care.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Healthcare use | 6 months
  Data on the changes in healthcare use will be collected from medical records

SECONDARY OUTCOMES:
Clinical impact and acceptability | 12 months post initiation of hypoallergenic formula containing synbiotics
  Clinical outcomes related to CMA and parent/carer and infant acceptability will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Nutricia UK
Locations (1):
- Adam Practice, Poole, United Kingdom

IPD SHARING:
Plan to Share IPD: No